CLINICAL TRIAL: NCT02781623
Title: Quantifying Quadriceps Atrophy Following Tibial Plateau Fracture
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: 15-00985
Record Dates: First submitted 2016-05-20; First posted 2016-05-24 (Estimated); Last update posted 2022-11-16 (Actual); Status verified 2022-11

CONDITIONS: Atrophy
Keywords: Quadriceps; Tibial Plateau; Fracture
MeSH Terms: conditions — Atrophy; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- MRI: An MRI will be conducted pre-operatively, 3 months post-operatively, and 1 year post-operatively.
  Interventions: Procedure: MRI

INTERVENTIONS:
Procedure: MRI

SUMMARY:
This study will quantify and examine the extent to which the quadriceps femoris muscle group atrophies following tibial plateau fractures and the length of time that atrophy affects function. The study will also look at the effects of tibial plateau fractures on the quadriceps muscle and the effect this atrophy has on functional outcome. Quadriceps atrophy will be measured both clinically and by using MRI scans taken pre-operatively, 3 months post operatively, and 1 year post-operatively. The injured leg and the non-injured leg will be scanned in order for the non-injured leg to serve as the control. In this way muscle volume can be estimated from the muscle thickness at specific locations in the thigh. The muscle strength of the quadriceps will also be assessed at the 3 month and 1 year visit by measuring isokinetic knee-extension torque, and functional assessment questionnaires will be completed at each study visit.

ELIGIBILITY:
Inclusion Criteria:

* All racial and ethnic groups
* Diagnosis of tibial plateau fracture
* Patients who opt for surgical treatment or non-operative treatment of their fracture
* Patients who consent to undergoing 3 MRI scans
* Patients who are willing to follow-up for a minimum of 52 weeks

Exclusion Criteria:

* Patients younger than 18 years old or older than 65
* Patients who may be pregnant or may become pregnant in the 52 weeks following injury
* Patients who have electric, magnetic, or mechanical devices currently implanted
* Patients who have abnormal ECG results
* Diagnosis of any additional lower extremity fractures other than tibial plateau
* Patients who fit the definition of a vulnerable population

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who opt for surgical treatment or non-operative treatment of their fracture.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2022-01-18 (Actual)

PRIMARY OUTCOMES:
Cross-sectional area (CSA) calculations | 1 Year
  From the axial images obtained from the MRI for each leg, outlines of each muscle in the quadriceps femoris muscle group will be traced and used to calculate.
Quadriceps muscle strength | One Year
  This will be measured by the highest knee-extension torque over six repetitions for each leg.
Muscle Volume | One Year
  This will be measured by the sum of the CSAs (Cross Sectional Areas) of each image times the thickness (10mm) and interslice gap (10mm) of each section
Pain Level | One Year
  This will be measured by the Short Musculoskeletal Function Assessment Questionnaire (SMFA)

SECONDARY OUTCOMES:
Isokinetic Knee-Extension Strength Test | One year
  This test will be conducted on both legs to compare the physical strength of the injured leg with the non-injured leg.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneeth Egol, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University Langone Medical Center, New York, New York, United States